CLINICAL TRIAL: NCT03691467
Title: The Effect of Hyaluronic Acid on Implant Stability After Immediate Implant Placement in Anterior and Premolar Region in Systemically Healthy Patients
Brief Title: the Effect of Topical Application of Hyaluronic Acid on Immediate Dental Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ibrahim Samy Kalboush (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Ibrahim Samy Kalboush, Associate lecturer in periodontology and oral medicine department Delta University, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: perio1088
Record Dates: First submitted 2018-09-28; First posted 2018-10-01 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Immediate Dental Implant
Keywords: immediate dental implant; immediate implant; hyaluronic acid; gengigel
MeSH Terms: interventions — Immediate Dental Implant Loading; Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Participant, Investigator
Masking Description: by addition of placebo gel in the control group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- immediate implant with hyaluronic acid. (Experimental): immediate dental implant with topical application of hyaluronic acid.
  Interventions: Device: immediate dental implant; Drug: Hyaluronic Acid
- immediate implant. (Active Comparator): immediate dental implant placement with placebo gel
  Interventions: Device: immediate dental implant

INTERVENTIONS:
Device: immediate dental implant — immediate dental implant placement in freshly extracted socket.
  Other Names: post extraction dental implant
Drug: Hyaluronic Acid — topical application of hyaluronic acid
  Other Names: gengigel
  Arms: immediate implant with hyaluronic acid.

SUMMARY:
The high predictability of immediate dental implants has led to routine use with a great expectation for success.

Immediate implant placement in fresh extraction sockets was reported to reduce alveolar bone resorption, Better esthetic outcomes were achieved including the prosthetic crown length in harmony with the adjacent teeth, natural scalloping and easier distinct papillae to achieve and maximum soft tissue support.

hyaluronic acid can be placed in freshly extracted sockets immediately after tooth extraction , also it could be used on implant surface in which hyaluronic acid enhance new bone formation around dental implants.

DETAILED DESCRIPTION:
Immediate dental implant placement was introduced more than 30 years ago by Schulte and Heimke in 1976.

The major advantages of immediate implant placement are reduction in number of visits, thus reduces the treatment time and improves patient satisfaction, provides ideal three dimensional implant position, and preserves the alveolar bone in the extraction socket

. However, immediate implants may have some disadvantages that can affect the success rate, which include inadequate primary implant stability when compared with delayed implants, inadequate soft tissue closure especially in case of thin tissue biotype, inability to inspect all aspects of the extraction site for defects or infection, and finally the added cost of bone grafting when the jumping distance is over 2mm.

Hyaluronic acid (HA) is one of the extracellular components of the connective tissue that belongs to the family of glycosaminoglycans, due to its non-immunogenic and non-toxic properties , it can be used in many medical fields such as dentistry, ophthalmology, dermatology.

HA has an important role in wound healing through inducing early granulation tissue formation, inhibiting destructive inﬂammatory process during the process of tissue healing, inducing re-epithelialization and angiogenesis.

HA not only acted as a carrier of growth factors and cells but also stimulated bone formation through chemotaxis, proliferation and differentiation of mesenchymal cells into osteoblasts. Although HA shares bone induction properties with osteogenic growth factors as bone morphogenic protein 2 and osteopontin.

HA also has anti-inflammatory effect through scavenging reactive oxygen species, such as superoxide radical (O2) and hydroxyl radical (OH) species, and inhibiting neutrophil derived serine proteinases, HA also has anti-edematous effect that may be related to its osmotic buffering capacity.

So surrounding of an implant with hyaluronic acid give a great potential to improve new bone formation and improve bone/implant contact which will improve healing time and implant stability.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients indicated for single or multiple immediate implants in anterior and premolar region. Absence of any peri-apical pathosis. Patients with intact buccal plate of bone. Patients with adequate bone volume for the dental implant procedure. Patient consent approval and signing.

Exclusion Criteria:

* Smokers. Systemic disease that may affect the final outcome of the surgical procedure. No or poor patient's compliance. Patients with psychological problems. Pathology at the site of intervention. Pregnant patients. Patients refuse to sign an informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
implant stability | 6 months
  implant stability using osstell "implant stability quotient (ISQ)"

SECONDARY OUTCOMES:
soft tissue healing | 10 days
  assessment of soft tissue healing using likert scale from (0-4) with 0: Complete wound closure without presence of fibrin and 4:Incomplete wound closure (necrosis).
post operative pain | 0-2 and 7 days
  assessment of pain severity with 10 point visual analogue scale (VAS) no pain '0' to severe/unbearable pain '10'

CONTACTS AND LOCATIONS:
Overall Officials: Mona shoeib, Doctor's, Study Chair — Cairo University; Mona Darhous, Doctor's, Study Chair — Cairo University
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
i will check with my study chair

REFERENCES:
- [Background] Schulz MC, Korn P, Stadlinger B, Range U, Moller S, Becher J, Schnabelrauch M, Mai R, Scharnweber D, Eckelt U, Hintze V. Coating with artificial matrices from collagen and sulfated hyaluronan influences the osseointegration of dental implants. J Mater Sci Mater Med. 2014 Jan;25(1):247-58. doi: 10.1007/s10856-013-5066-3. Epub 2013 Oct 11. PMID 24113890
- [Background] Lee JH, Kim J, Baek HR, Lee KM, Seo JH, Lee HK, Lee AY, Zheng GB, Chang BS, Lee CK. Fabrication of an rhBMP-2 loaded porous beta-TCP microsphere-hyaluronic acid-based powder gel composite and evaluation of implant osseointegration. J Mater Sci Mater Med. 2014 Sep;25(9):2141-51. doi: 10.1007/s10856-014-5250-0. Epub 2014 Jun 14. PMID 24928668